CLINICAL TRIAL: NCT06157463
Title: 68Ga FAPI in Total Neoadjuvant Therapy of Rectal Cancer
Brief Title: FAPI in Rectal Cancer TNT
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 202202030A0C601
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-11

CONDITIONS: Rectal Neoplasms Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation: Ga-68 FAPI study before and during TNT
  Interventions: Radiation: Ga-68 FAPI

INTERVENTIONS:
Radiation: Ga-68 FAPI — FAPI PET scans will be performed in addition to other staging/restaging work-up

SUMMARY:
The goal of the trial is to observe the changes of 68Ga FAPI signal before and after total neoadjuvant therapy for rectal cancers, and the correlation between the image parameters, immune checkpoints expression as well as the patient outcome. The trial will recruit patients with biopsy-confirmed rectal cancer aged 18 years old or older, with WHO/ECOG Performance Status 0-1, and eligible for total neoadjuvant therapy at the clinicians' discretion. After signing the informed consent, the participants will undergo a standard staging work-up if not already done, including colonoscopy and cross-sectional images such as CT, MR, and FDG-PET. Kidney function (by serum creatinine) and liver function (by serum alanine aminotransferase) will also be assessed. Only patients with stage II-III rectal cancer will be recruited.

If patients meet the inclusion and exclusion criteria, they will undergo the first 68Ga-FAPI PET within 30 days before the beginning of total neoadjuvant therapy. At 22-24 weeks into the TNT, follow-ups for response evaluation will be conducted, including colonoscopy and cross-sectional images such as CT, MR, and FDG-PET. The second 68Ga-FAPI PET will be performed within one month of these exams. Afterward, participants will either undergo surgery or have image follow-ups every 3 months. The participants will be followed up for up to 2 years after the second 68Ga-FAPI PET, and immunochemical staining with CD47, CD73, PD-L1, and FAP on the biopsy or surgical specimens will be performed in one batch to avoid batch-to-batch variation.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven newly detected adenocarcinoma of the rectum
2. Clinical stage II-III rectal cancer
3. Aged at least 18 years. No upper age limit.
4. WHO/ECOG Performance Status 0-1
5. Eligible for total neoadjuvant therapy

Exclusion Criteria:

1. Distant metastases found on either CT, MR or FDG-PET
2. Prior anticancer therapy for colorectal cancer
3. Prior radiotherapy of the pelvic region
4. Other concurrent antineoplastic therapy
5. Major surgery within the last 4 weeks prior to inclusion
6. Subjects pregnant or breast feeding
7. Serious concurrent diseases not compatible with study entry, including active, uncontrolled infections, active, disseminated coagulation disorder, clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia within 6 months before enrolment)
8. Neurologic or psychiatric disorders including dementia, uncontrolled seizures, substance abuses, severe depression
9. Prior or concurrent malignancy within 3 years prior to enrolment (except non-melanoma skin cancer or cervical carcinoma FIGO stage 0-1)
10. Allergic to contrast agents or to the main ingredients or excipients of the experimental radiopharmaceutical 68Ga FAPI, including acetate, ascorbic acid and normal saline
11. Those deemed unsuitable for participation in the trial by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those patient referred to the tertiary medical center for rectal cancer will be invited to enroll in the study.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of FAPI SUV | before TNT & 22-24wk into TNT
  To compare the FAPI uptake after TNT

SECONDARY OUTCOMES:
Correlation of FAPI SUV | 2 years after recruitment
  FAPI SUV will be correlated with (1) 2-year disease-free survival (DFS), (2) 2-year local regional recurrence (LRR), (3) 2-year total mesorectal excision (TME)-free survival, (4) 2-year overall survival (OS), (5) overall complete response (CR) rate, and (6) immune checkpoint protein expression including CD47, CD73, PD-L1, and FAP

CONTACTS AND LOCATIONS:
Overall Officials: Shih-hsin Chen, MD PhD, Principal Investigator — Chang Gung Medical Foundation
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared with co-investigators listed in the IRB application to protect the participants' privacy.